CLINICAL TRIAL: NCT06191614
Title: Multi-center, Single-group, Prospective Observational Study to Evaluate the Efficacy of DEXINEURO Tab on Blood Glucose Reduction in Type 2 Diabetic Patients With Diabetic Peripheral Neuropathy
Brief Title: DEXINEURO® Tab on Blood Glucose Reduction in Patients With Type 2 Diabetes Accompanied by Diabetic Peripheral Neuropathy
Status: Completed | Type: Observational
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: HL-DXNR-401
Record Dates: First submitted 2023-12-17; First posted 2024-01-05 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: R-thioctic acid tromethamine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to evaluate the efficacy of DEXINEURO® tab on blood glucose reduction and assess the interaction with concomitantly administered insulin or oral antidiabetic agents in patients with type 2 diabetes accompanied by diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
This clinical trial is a multi-center, single-group, prospective observational study conducted to investigate the interaction with concomitant insulin or oral antidiabetic agents and assess the influence on blood glucose reduction when administering DEXINEURO® tab to patients with type 2 diabetes and diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years and older of both genders.
2. Type 2 diabetes patients with HbA1c ≤ 10% at screening.
3. Patients diagnosed with diabetic peripheral neuropathy who are scheduled to receive DEXINEURO® tab.
4. Individuals who have voluntarily provided written consent to participate in this study.

Exclusion Criteria:

1. Individuals who have taken or are currently taking alpha-lipoic acid (thioctic acid) within 1 month before screening.
2. Individuals contraindicated according to the approval conditions of DEXINEURO® tab.
3. Pregnant or breastfeeding women.
4. Individuals participating in other clinical trials (except for non-interventional observational studies, if they have not received investigational drugs, or are participating in other non-interventional observational studies).
5. Individuals whom the principal investigator deems inappropriate for participation in this study for reasons other than those mentioned above.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Prescribed DEXINEURO® tab for the treatment of diabetic peripheral neuropathy
Sampling Method: Probability Sample
Enrollment: 528 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in fasting plasma glucose (FPG) after 12 of DEXINEURO® tab administration compared to baseline | after 12 weeks of prescription for DEXINEURO tab compared to baseline
  Change in fasting plasma glucose (FPG) after 12 of DEXINEURO® tab administration compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ho-chan Cho, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (1):
- Keimyung University Dongsan Hospital, Daegu, South Korea